CLINICAL TRIAL: NCT04762238
Title: Does the Diacutaneous Fibrolysis Change Ultrasonographic Measurements in Patients With Carpal Tunnel Syndrome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sandra Jiménez, PhD Physiotherapist, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Zaragoza
Record Dates: First submitted 2021-02-10; First posted 2021-02-21 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Carpal Tunnel Syndrome; Physical Therapy Modalities; Ultrasonography
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual Diacutaneous Fibrolysis (Experimental): Diacutaneous Fibrolysis is a non invasive physiotherapeutic technique applied by means of a set of metallic hooks ending a spatula with bevelled edges that help to treat the muscles and conjunctive tissues and trying to improve mobility between mobility between muscle planes.
  Interventions: Other: Diacutaneous Fibrolysis
- Sham Diacutaneous Fibrolysis (Sham Comparator): Sham Diacutaneous Fibrolysis is applied at a superficial level. A pinch of skin was held with the thumb of the palpatory hand and the tip of the spatula but without effect in the muscle because no penetrate in deep tissue
  Interventions: Other: Diacutaneous Fibrolysis

INTERVENTIONS:
Other: Diacutaneous Fibrolysis — Diacutaneous Fibrolysis is a non invasive physiotherapeutic technique applied by means of a set of metallic hooks ending a spatula with bevelled edges that help to treat the muscles and conjunctive tissues and trying to improve mobility between mobility between muscle planes.

SUMMARY:
The carpal tunnel syndrome (CTS) is a common entrapment neuropathy caused by compression of the median nerve at the wrist.Clinically electroneuphysiological assessment is not accessible to all clinicians. In this way ultrasounds (US) is a more accessible and economical tool and many studies have reported that US has high sensitivity and specificity in the diagnosis of CTS.Diacutaneous Fibrolysis (DF) is a physiotherapeutic technique derived from Cyriax deep friction massage principles.DF technique could assist in improving changes in the connective tissues adjacent to the median nerve, especially the thickness of TCL and this could be reflected in a decreasing of TCL. Moreover, the neurophysiological and mechanical effect described by this technique may improve the nerve compression decreasing the CSA of the median nerve.

The purpose of this study is to quantify changes in the cross-sectional area of the median nerve in the carpal tunnel and the thickness of transversal carpal ligament measured by US and the changes in the intensity of the numbness and the subjective assessment of clinical change after DF treatment in forearm, wrist and hand area compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed medically with neurophysiological test of carpal tunnel syndrome (low and moderate intensity)

Exclusion Criteria:

* Severe carpal tunnel syndrome
* Previous surgery on the hand
* hormonal factors: diabetes, thyroids pathologies, pregnant
* Cervical disfunctions
* Ulcerations or skins disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Cross sectional area of the median nerve with ultrasonography | Baseline (Before the treatment)
  Cross sectional area of the median nerve with ultrasonography at carpal tunnel level
Cross sectional area of the median nerve with ultrasonography | After treatment application, an average of 2 weeks
  Cross sectional area of the median nerve with ultrasonography at carpal tunnel level

SECONDARY OUTCOMES:
Intensity of numbness with the Visual Analogue Scale (VAS 1-10cm) | Baseline (Before the treatment)
  Intensity of numbness with Visual Analogue Scale (1-10cm)
Intensity of numbness with the Visual Analogue Scale (VAS 1-10cm) | After treatment application, an average of 2 weeks
  Intensity of numbness with Visual Analogue Scale (1-10cm)
Thicknesses of transverse carpal ligament with ultrasonography | Baseline (Before the treatment)
  the thicknesses of transverse carpal ligament on the cross-section at the level of hamate bone with ultrasonography at carpal tunnel level
Thicknesses of transverse carpal ligament with ultrasonography | After treatment application, an average of 2 weeks
  the thicknesses of transverse carpal ligament on the cross-section at the level of hamate bone with ultrasonography at carpal tunnel level
Subjective assessment of clinical change with the Global Rating of Change Scale (GROC Scale) | After treatment application, an average of 2 weeks
  Subjective assessment of clinical change with Global Rating of Change Scale (GROC scale) a scale ranging from -7 ("a very great deal worse") to 0 ("about the same") to +7 ("a very great deal better").

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jiménez-del-Barrio, PhD, Principal Investigator — University of Valladolid
Locations (1):
- Sandra Jiménez Jiménez-del-Barrio, Soria, Spain

IPD SHARING:
Plan to Share IPD: No